CLINICAL TRIAL: NCT05325372
Title: A Comparative Study Between the Ultrasound-guided Infraclavicular Block and Axillary Block for Assessment of Motor Power Degree and Duration Using Handgrip Dynamometer in Patients Undergoing Minor Hand Surgery. A Randomized Control Trial
Brief Title: A Comparative Study Between Infraclavicular and Axillary Blocks for Assessment of Motor Power Using Handgrip Dynamometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Lecturer of anesthesia (principal investigator), Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-529-2021
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Hand Surgery; Ultrasound Guided

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer-generated numbers and concealed by serially numbered, opaque, and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in a set of sealed envelopes each bearing only the case number on the outside.
  This study will be performed by 3 anesthetists; one anesthetist who is experienced in performing the blocks will be allocated to perform either the axillary or infraclavicular block according to a computer-generated sequence of random numbers and sealed envelope, and the other two anesthetists will be blinded to the technique performed, and they will monitor the patients intra and postoperatively. Assessment of brachial plexus blockade will be carried out every 10 mins until 30 min by one of these two blinded observers. The infraclavicular and axillary areas will be covered to maintain the blinding of investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided axillary block (Experimental): the Ultrasound probe with a linear high frequency (8-14 MHZ) transducer will be placed parallel to the anterior axillary fold at the axilla to identify the axillary artery and to identify the hyperechoic median, ulnar, and radial nerves in relation to the axillary artery. The musculocutaneous nerve which supplies the skin of the lateral side of the forearm had to be blocked also. It is found between the biceps brachii and coracobrachialis muscles. Lidocaine 1% was infiltrated subcutaneously 1 cm lateral to the probe. The needle is inserted in-plane from the anterior aspect and directed toward the posterior aspect of the axillary artery. All four nerves in the axillary region will be blocked. A local anesthetic will be administered adjacent to each of the four nerves (at least 5 ml for each).
  Interventions: Procedure: axillary block
- Ultrasound guided infraclavicular block block (Experimental): The transducer is positioned in the parasagittal plane to identify the axillary artery. Surrounding the artery are the three cords of the brachial plexus: the lateral, posterior, and medial cords. The needle is inserted in-plane short-axis technique from the cephalad end of the probe, with the insertion point just inferior to the clavicle. A local anesthetic will be injected posterior to the axillary artery to achieve a U-shaped distribution around the artery (cephalad, caudad, and posterior).
  Interventions: Procedure: infraclavicular block

INTERVENTIONS:
Procedure: axillary block — it will be given using 20 ml of drug 0.25% bupivacaine (10 ml 0.5% bupivacaine + 10 ml normal saline).
  Other Names: peripheral nerve block
  Arms: Ultrasound guided axillary block
Procedure: infraclavicular block — it will be given using 20 ml of drug 0.25% bupivacaine (10 ml 0.5% bupivacaine + 10 ml normal saline).
  Other Names: peripheral nerve block
  Arms: Ultrasound guided infraclavicular block block

SUMMARY:
Hand Surgery is surgery of the hand, the wrist, and the peripheral nerves of the upper limb. Many different types of surgeries can be performed on the hand, depending on the underlying cause of the problem such as Closed reduction and fixation, Tendon repair, Skin grafts, Skin flaps, Carpal Tunnel Release, and ganglion removal. Hand surgery is usually associated with marked postoperative pain. Ultrasound-guided regional anesthesia is usually performed in patients undergoing hand surgery.

This study aims to compare Ultrasound-guided infraclavicular block and axillary block and assess the degree of motor power and duration by testing hand grip strength using a hydraulic hand dynamometer in patients undergoing hand surgery.

Objectives:

To determine the degree of a motor block using a hydraulic hand dynamometer. To Estimate time needed to regain full motor activity. To identify whether ultrasound-guided axillary block may preserve motor function to a greater extent than infraclavicular blocks.

DETAILED DESCRIPTION:
This randomized control trial is designed to include (52) patients ASA physical status I, II patients ranging from(18) to(60)years old scheduled for hand surgery

Patients meeting the inclusion criteria will be randomly assigned to receive either:

Group I: axillary block technique (n=26) (group A) GroupII: infraclavicular block technique( n=26)(group B) Anesthesia management After arrival to the anesthetic room, An 18-gauge intravenous cannula will be placed at the forearm contralateral to the operated arm, standard monitoring will be used (non-invasive arterial blood pressure, ECG, pulse oximetry) while performing the block and throughout the surgical procedure. Premedication will be given intravenously in the form of 0.03 mg/kg midazolam. 1 g paracetamol iv will be given for all patients Under aseptic conditions, a preliminary scan will be performed using siemens acuson x 300 ultrasound with 8-14 MHz linear transducer. A 50-mm block needle 22 gauge will be used. (SonoPlex Stim Cannula, Germany) All blocks will be given by one researcher using 20 ml of drug 0.25% bupivacaine (10 ml 0.5% bupivacaine + 10 ml normal saline).

Axillary block

Patients in group A will be placed in the supine position with the arm to be blocked abducted and externally rotated. After sterilization of the axilla, the Ultrasound probe with a linear high frequency (8-14 MHZ) transducer will be placed parallel to the anterior axillary fold at the axilla to identify the axillary artery and to identify the hyperechoic median, ulnar, and radial nerves in relation to the axillary artery. The musculocutaneous nerve which supplies the skin of the lateral side of the forearm had to be blocked also. It is found between the biceps brachii and coracobrachialis muscles. Lidocaine 1% was infiltrated subcutaneously 1 cm lateral to the probe. The needle is inserted in-plane from the anterior aspect and directed toward the posterior aspect of the axillary artery. All four nerves in the axillary region will be blocked. A local anesthetic will be administered adjacent to each of the four nerves (at least 5 ml for each).

Infraclavicular block

Patients in group B will be placed in the supine position with the head turned away from the side to be blocked. The arm is abducted to 90 degrees and the elbow flexed. the skin is disinfected and the transducer is positioned in the parasagittal plane to identify the axillary artery. Surrounding the artery are the three cords of the brachial plexus: the lateral, posterior, and medial cords. The needle is inserted in-plane short-axis technique from the cephalad end of the probe, with the insertion point just inferior to the clavicle. A local anesthetic will be injected posterior to the axillary artery to achieve a U-shaped distribution around the artery (cephalad, caudad, and posterior).

Injection of 5 ml lidocaine 2% will be also used in all patients to eliminate tourniquet pain and pain in the area of distribution of intercostobrachial nerve in case of use of a tourniquet

Block assessment

After completion of all block procedures. A formal assessment of block efficacy will be performed by an independent observer who will be masked to each subject's group allocation every 10 min after needle removal for 30 min. surgery will be started once surgical anesthesia will be achieved at any time point or until 30 min had elapsed. if surgical anesthesia will not be achieved at 30 min the block will be considered failed and general anesthesia will proceed.

Sensory blockade of the musculocutaneous, median, radial and ulnar nerves will be graded according to the previously validated 3 point scale using a cold test: respectively: 0 = no perception, 1 = decreased sensation, or 2 = normal sensation. A successful blockade is defined as a complete sensory blockade (i.e., sensory block score = 0) within 30 minutes of completing the block. If complete sensory blockade will not be achieved within 30 minutes, the affected subject will be excluded from the study and categorized as a block failure. The subject was offered a supplementary nerve block if there is sufficient time before surgery, or general anesthesia will be proceeded to achieve surgical anesthesia.

The procedural time (seconds) for each block will be recorded. This duration is defined as the interval from the ultrasound transducer's first contact with the subject to the time the block needle exit the skin. Block onset time will be recorded (from a completed injection of local anesthetic until loss of cold sensation) Duration of the block will be recorded, defined as the time from completing injection of the local anesthetic till complete recovery of sensory function, i.e., the cold test will be assessed every 30 min in the postoperative period till patient feel the cold sensation

The motor blockade will be assessed by testing patients' handgrip strength using a hydraulic handgrip dynamometer, baseline measurements will be recorded on both the ipsilateral and contralateral sides. hand grip strength will be measured preoperative, 30 min from a block, and after surgery. postoperative change in handgrip strength in the operative limb as a percent reduction of preoperative baseline strength will be measured. The time needed to regain full motor power will be measured.

All patients will be postoperatively monitored in the post-anesthesia care unit (PACU) for 1 h and thereafter discharged to their wards. Post-operative pain at the incision site will be assessed by visual analog scale (VAS) and a score of more than 3 when recorded will be taken as an endpoint for the duration of block and the patient was given supplementary analgesics i.e. Inj. Diclofenac Sodium 1-1.5 mg/kg intramuscular. Subject satisfaction will be assessed with a standardized question scored on a seven-point Likert scale: "Thinking about your nerve blocks, how satisfied were you with them: where 1 is not at all, 4 is neutral, and 7 is completely satisfied?"

Block related complications will be recorded such as failed block, motor weakness 24 h after the block local anesthetic toxicity, vascular puncture, paraesthesia, and pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

1. Gender both males and females
2. ASA Class I, II
3. Age 18-60 years
4. Patients undergoing minor hand surgery (skin graft, Carpal Tunnel Release, ganglion removal, and lipoma ) expected surgical time of more than 15 min and less than one hour.

Exclusion Criteria:

1. Allergy to local anesthetic
2. Infection of the skin at the site of block.
3. Bilateral surgery, neck and clavicle deformities, existing neurological disease chronic pain diagnosis, pre-existing nerve damage, muscle injuries, and tendon injury.
4. Coagulopathy, previous surgery on the operative limb, inability to comprehend study-related procedures, and clinically significant cognitive impairment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Postoperative change in handgrip strength in the operative limb | it will be measured at 90 min from the block
  Postoperative change in handgrip strength in the operative limb as a percent reduction of preoperative baseline strength at 90 min from the block (%)

SECONDARY OUTCOMES:
Block related complications | it will be measured in the first 24 hours postoperative
  local anesthetic toxicity, vascular puncture, paresthesia, and pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Yasser EL Halafawy, professor, Study Director — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No